CLINICAL TRIAL: NCT02777879
Title: Lung Microbiome and Inflammation in Early Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Lung Microbiome and Inflammation in Early COPD
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01546
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstuctive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Microbial DNA will be extracted from sputum and BAL fluid. Variable 16S rRNA gene regions will be amplified by PCR using bar-coded primers flanking a portion of marker gene. PCR products will be sequenced in the NYU Genome Technology Center using MiSeq platform (Illumina).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Obstructive Pulmonary Disease (COPD): Case of early COPD (GOLD 1-2, FEV1/FVC<70 and FEV1>50%)
  Interventions: Procedure: Bronchoscopy
- Control: No obstruction (FEV1/FVC<70). Controls will be recruited after each case and will be matched by: age (±5 year), 2) gender, 3) smoking (±5 pack-year) and 4) BMI (±5).
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Flexible bronchoscopy with bronchoalveolar lavage (BAL) and bronchial brushings will be done in a standardized manner. The bronchoscope tip is sequentially wedged in sub-segments where BAL will be performed on a total of two segments of the lung (120 ml in each segment for a total of 360 ml). Two brushes will be done under direct visualization in both segments. Selection of segments to sample will be based on where abnormalities are in imaging.

SUMMARY:
This is a cross sectional case controlled study to assess lung microbiome and inflammation in smokers with and without Chronic Obstructive Pulmonary Disease (COPD). Investigators will look at active bacterial metabolic pathways in the lower airways using metagenomic and metabolomic approaches an assess relationships among microbiome, metagenome, metabolome and host immune responses in COPD and controls. Investigators believe COPD cases will have higher prevalence of pneumotype supraglottic predominant taxa (SPT) than matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Case definition: Smokers (>20 pack-year) with airflow obstruction (FEV1/FVC<70) and FEV1>50% predicted (early COPD GOLD 1 or 2)
* Control definition: Smokers with normal spirometry will serve as controls.

Exclusion Criteria:

* FEV1 < 50% NOT 70
* Significant cardiovascular disease defined as abnormal EKG, known or suspected coronary artery disease or congestive heart failure.
* Diabetes mellitus
* Significant liver or renal disease
* Severe coagulopathy (INR > 1.4, PTT > 40 seconds and platelet count < 150x103 cells).
* Pregnancy
* ETOH use of more than >6 beers or >4 mixed drinks daily
* Lack of capacity to provide informed consent.
* Antibiotic use within the prior 2months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Utilizing cohorts built at NYU over the last several years, this project is uniquely positioned to investigate the microbiome signatures among subjects with COPD.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2014-05; Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Site specific microbiome (supraglotic area) constituents using background subtraction and source tracking approaches via a multivariable conditional logistic regression model. following broncho-alveolar lavage, BAL | 4 Hours

SECONDARY OUTCOMES:
Bacterial metabolic pathways in the lower airways using metagenomic and metabolomic approaches | 4 Hours
  Bioinformatic methods such as Procrustes will be used to integrate the analysis of the generated multi-omic datasets through this study to attain a more accurately defined COPD phenotype. By elucidating the interplay between bacterial composition, microbiome functional repertoire, metabolism, and immunological status in the human lung, we will obtain further insights for hypothesis generation into the pathophysiological mechanisms underlying COPD.

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Segal, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States